CLINICAL TRIAL: NCT01045863
Title: A Phase 1, First-Into-Human, Escalating Dose Trial To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of PF-03382792 After Administration Of Single Oral Doses To Healthy Adult Subjects
Brief Title: To Evaluate Safety, Tolerability, Plasma Drug Levels And Other Biological Effects In Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: B1651001
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PART A: Ascending Cohorts (Experimental): Single ascending dose cross-over. (0.05, 0.15, 0.5, 1.5, 5, 15 mg)
  Interventions: Drug: PF-03382792 Cohort 1; Drug: PF-03382792 Cohort 2; Drug: PF-03382792
- PART B: Food effect (Experimental): Food effect on PF-03382792 PK
  Interventions: Drug: Food Effect cohort
- PART C: CSF Cohort (Experimental): Optional CSF Cohort
  Interventions: Drug: CSF cohort

INTERVENTIONS:
Drug: PF-03382792 Cohort 1 — First cohort for: Single oral ascending dose of PF-03382792, formulated in solution.
  Arms: PART A: Ascending Cohorts
Drug: PF-03382792 Cohort 2 — Second cohort for: Single oral ascending dose of PF-03382792, formulated in solution.
  Arms: PART A: Ascending Cohorts
Drug: PF-03382792 — Optional cohort 3: Single oral ascending dose of PF-03382792, formulated in solution.
  Arms: PART A: Ascending Cohorts
Drug: Food Effect cohort — Single oral dose, cross-over to determine effect of food on PF-03382792 pharmacokinetics. Dose will be decided after reviewing data from the ascending dose portion.
  Arms: PART B: Food effect
Drug: CSF cohort — Single oral dose of PF-03382792 formulated in solution. Dose will be decided after reviewing data from the ascending dose portion.
  Arms: PART C: CSF Cohort

SUMMARY:
The purpose of this study is to evaluate safety and tolerability after a single administration of PF-03382792 in healthy volunteers.; and to evaluate plasma drug levels and biological activity.

DETAILED DESCRIPTION:
Evaluate the safety, tolerability, plasma concentrations of PF-03382792 and other biological activity following a single dose of PF-03382792. Three ascending single doses of PF-03382792 were administered in this study (0.05 mg, 0.15mg and 0.5 mg). The decision to terminate the study was made on June 4, 2010 due to safety findings and limitations regarding the levels of the metabolite projected for doses above 0.5 mg.

ELIGIBILITY:
Inclusion Criteria:

* For all cohorts, healthy male and/or female subjects of nonchildbearing potential between the ages of 18 and 55 years, inclusive.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* Signs or symptoms of adrenal insufficiency.
* Ocular lens (eye) abnormalities.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety endpoints include evaluation: adverse events, change from baseline in vital signs, triplicate ECG (Part A only), singlet ECG for Parts B and C. 8 hours of cardiac telemetry postdose (Part A only). | For cohorts in Part A, up to 24 days; for Cohorts in Part B, up to 17; for Part C, up to 10 days
Additional Safety endpoints: clinical safety laboratory endpoints, plasma cortisol and ACTH, clinical examinations, slit lamp examination. | For cohorts in Part A, up to 24 days; for Cohorts in Part B, up to 17; for Part C, up to 10 days
Pharmacokinetic endpoints: plasma concentration of PF 03382792 over time (eg, AUC, Cmax, Tmax, t1/2), plasma concentration of PF 03227077 over time (eg, AUC, Cmax, Tmax, t1/2). | up to 72 hours post the final dose for each cohort

SECONDARY OUTCOMES:
Plasma aldosterone concentrations. | For Part A and C; up to 24 hours post final dose
Change and percent change from baseline in average CSF sAPP fragment concentrations over all postdose collection time points up to 8 hours. • CSF sAPP fragment concentrations over time. • CSF concentration of PF 03382792 and PF | Part C only, up to 8 hours post dose
03227077 over time (eg, AUC, Cmax, Tmax). | Part C only, up to 8 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1651001&StudyName=To%20Evaluate%20Safety%2C%20Tolerability%2C%20Plasma%20Drug%20Levels%20And%20Other%20Biological%20Effects%20In%20Healthy%20Volunteers